CLINICAL TRIAL: NCT02788435
Title: The Role of Voice Rest on Voice Outcomes Following Phonosurgery: A Randomized-Controlled Trial
Brief Title: The Role of Voice Rest on Voice Outcomes Following Phonosurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107893
Record Dates: First submitted 2016-05-16; First posted 2016-06-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Unilateral Vocal Cord Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients in the control arm will undergo a graduated prescription of voice use immediately following surgery.
- Absolute Voice Rest (Experimental): Patients in the experimental arm will undergo 7 days of absolute voice rest following surgery.
  Interventions: Behavioral: Absolute Voice Rest

INTERVENTIONS:
Behavioral: Absolute Voice Rest — Patients will be instructed to not use their voice and minimize any voice-use activities such as coughing or throat-clearing for a period of 7 days following surgery.
  Arms: Absolute Voice Rest

SUMMARY:
Patients undergoing vocal cord surgery (phonosurgery) are often prescribed voice rest postoperatively. However, no clinical trials have ever been conducted to ascertain the efficacy of using voice rest and its impact on functional voice outcomes. The purpose of this randomized-clinical trial is to determine if the prescription of voice rest has an impact on voice outcomes following phonosurgery.

DETAILED DESCRIPTION:
The study will seek to determine if a 7-day period of absolute voice rest alters voice-related quality of life following phonosurgery

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Unilateral vocal cord lesion
* Consented for phonosurgery

Exclusion Criteria:

* Age less than 18 years
* Bilateral vocal cord lesions
* Prior vocal cord surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index (VHI)-10 | 4 weeks post-operative
Voice Handicap Index (VHI)-10 | 12 weeks post-operative

SECONDARY OUTCOMES:
Frequency perturbation (jitter) | 4 weeks post-operative
Frequency perturbation (jitter) | 12 weeks post-operative
Amplitude perturbation (shimmer) | 4 weeks post-operative
Amplitude perturbation (shimmer) | 12 weeks post-operative
Fundamental frequency | 4 weeks post-operative
Fundamental frequency | 12 weeks post-operative
Maximum phonation time | 4 weeks post-operative
Maximum phonation time | 12 weeks post-operative
Perceptual grading of voice using the Grade, Roughness, Breathiness, Asthenia, Strain, Instability (GRBASI)-scale | 4 weeks post-operative
Perceptual grading of voice using the Grade, Roughness, Breathiness, Asthenia, Strain, Instability (GRBASI)-scale | 12 weeks post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fung, MD, FRCSC, Principal Investigator — Department of Otolaryngology - Head & Neck Surgery, Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhaliwal SS, Doyle PC, Failla S, Hawkins S, Fung K. Role of voice rest following laser resection of vocal fold lesions: A randomized controlled trial. Laryngoscope. 2020 Jul;130(7):1750-1755. doi: 10.1002/lary.28287. Epub 2019 Sep 9. PMID 31498467